CLINICAL TRIAL: NCT05089643
Title: Anrotinib in Combination With Capecitabine in the Single-arm, Open Phase II Treatment of Relapsed or Metastatic Triple-negative Breast Cancer Clinical Research
Brief Title: Anrotinib in Combination With Capecitabine in Advanced Triple Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Chief of VIP department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC1969
Record Dates: First submitted 2021-09-27; First posted 2021-10-22 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — anlotinib; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CA (Experimental): Anlotinib 10mg Qd D1-14 Capecitabine 1G /m2 Bid D1-14 / Q21D
  Interventions: Drug: Anlotinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Anlotinib — Before breakfast, anlotinib hydrochloride capsule was taken on an empty stomach, once a day, 1 tablet (10mg) each time.Continuous oral administration for 2 weeks stopped for 1 week, that is, 3 weeks (21 days) as a treatment cycle, until disease progression or adverse reactions become intolerable.In case of missing medication, confirm that the time before the next medication is less than 12 hours, no refill.
Drug: Capecitabine — Capecitabine tablets 1000 mg/m2, twice a day, within 30min after meals, were taken orally for 2 consecutive weeks and stopped for 1 week, i.e., 3 weeks (21 days) as a treatment cycle until disease progression or adverse reactions became intolerable.

SUMMARY:
The hypothesis of this study is to discover if the capecitabine plus Anlotinib can shrink or slow the growth of pretreated advanced TNBC.

It is a single-arm phase II clinical study of capecitabine combined with antinib in the treatment of recurrent or metastatic triple-negative breast cancer

DETAILED DESCRIPTION:
It is a single-arm phase II clinical study of capecitabine combined with antinib in the treatment of recurrent or metastatic triple-negative breast cancer.

The hypothesis of this study is to discover if the capecitabine plus Anlotinib can shrink or slow the growth of pretreated advanced TNBC.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged between 18 and 70;
2. Recurrence or metastasis OF TNBC confirmed by histological or cytological methods, TNBC definitions of ER, PR and HER-2 are negative, if there is metastasis pathology, the histological pathology of metastasis shall prevail.ER and PR negative were defined as ER < 10% positive and PR < 10% positive.
3. Disease progression after at least one prior systemic treatment and anthracycline and/or taxane use;Note: For neoadjuvant/adjuvant therapy, recurrence or disease progression during treatment or within 6 months of discontinuation of treatment should be counted as first-line systemic treatment failure;
4. There should be at least one measurable lesion according to the efficacy evaluation criteria for solid tumors (RECIST version 1.1)

Exclusion Criteria:

1. The number of previous treatment lines (including postoperative adjuvant therapy) >4 lines
2. symptomatic central system metastases.Patients with stable asymptomatic BMS who have received brain radiation and who have at least one other evaluable target in addition to the BMS can be enrolled (evaluable target should be at least 4 weeks away from the last radiotherapy).
3. New bisphosphonate or dinoselmer treatment for bone metastases was initiated within 28 days prior to study initiation.(Subjects are permitted if they have already been treated with bisphosphonate or dinoselmer for at least 4 weeks of optimal stable administration prior to study initiation.)Subjects already enrolled in this study may begin treatment with bisphosphonate or dinoselmer for bone metastases after the first post-treatment evaluation

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 1 year after the last patient enrolled
  he ORR will be defined as the proportion of patients in the Efficacy Evaluable patient Set who achieve complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Progression-free survival | up to 1 year after the last patient enrolled
  PFS will be defined as the time from first dose of study drug until documentation of disease progression or death from any cause
adverse events | approximately 1.5 years
  Incidence and Severity of adverse events hematologic，hepatotoxicity，Incidence of hypertension，Incidence of proteinuria

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing